CLINICAL TRIAL: NCT00673673
Title: Phase II Study of FOLFOX With Bevacizumab (Avastin(TM)) in Metastatic or Unresectable Gastroesophageal and Gastric Cancer
Brief Title: FOLFOX With Bevacizumab in Metastatic or Unresectable Gastroesophageal and Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0710003118
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Gastroesophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Folfox protocol; Oxaliplatin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): FOLFOX in combination with bevacizumab
  Interventions: Drug: FOLFOX; Drug: bevacizumab

INTERVENTIONS:
Drug: FOLFOX — Oxaliplatin 85/mg/m2 IV infused over two hours followed by Leucovorin 400 mg/m2 IV over 2 hours, followed by 5-FU 400 mg/m2 IV bolus, then 2400 mg/m2 continuous IV infusion over 46-48 hours
  Other Names: Eloxatin; Fluorouracil
Drug: bevacizumab — bevacizumab will be used at a dose of 10 mg/kg administered every 2 weeks on day one of FOLFOX chemotherapy
  Other Names: Avastin

SUMMARY:
This is a Phase II open-label study to determine the anti-tumor efficacy and tolerability of FOLFOX in combination with bevacizumab (Avastin(TM))in patients with metastatic or unresectable gastroesophageal and gastric adenocarcinoma. Our primary objective is to determine the time to progression in patients treated with FOLFOX in combination with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented recurrent, metastatic or unresectable gastroesophageal (Siewert type I, II, III) or gastric adenocarcinoma with measurable or assessable non-measurable disease (RECIST criteria).
* If recurrent or metastatic disease is not histologically confirmed, then documentation by a second radiographic procedure (i.e., PET scan or MRI in addition to CT scan) is required. If the imaging procedure does not confirm recurrent or metastatic disease, biopsy confirmation is required
* 12 months since completion of any prior neoadjuvant or adjuvant therapy (chemotherapy or radiotherapy) for potentially resectable gastroesophageal or gastric adenocarcinoma.
* >4 weeks since major surgery.
* ECOG Performance Status: 0-1
* Life expectancy >12 weeks
* Laboratory parameters as follows: absolute neutrophil count ≥1,500/uL, platelet count ≥100,000/uL, hemoglobin ≥9 g,/dL, creatinine <1.5 X ULN or estimated GFR >30 ml's/min, urinalysis <2+ protein, baseline proteinuria <1000 mg/d or urine protein/creatinine ratio <1, bilirubin <2 X ULN, PT (INR) <1.5 if patient not on anticoagulation, negative pregnancy test in women of childbearing age
* Hypertension must be well controlled (<160/90)
* Paraffin block or slides must be available
* Patients on full-dose anticoagulants must be on a stable dose of warfarin and have an in-range INR or be on a stable dose of low molecular weight heparin.

Exclusion Criteria:

* prior treatment for recurrent, metastatic, or unresectable gastroesophageal or gastric adenocarcinoma
* other concurrent anticancer therapy
* other malignancy within past three years except basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer known central nervous system metastases or carcinomatous meningitis.
* interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung.
* > grade 2 sensory peripheral neuropathy.
* uncontrolled seizure disorder, active neurological disease, or known CNS disease.
* significant cardiac disease, including the following: unstable angina, New York Heart Association class II-IV congestive heart failure, myocardial infarction within six months prior to study enrollment.
* history of hypertensive crisis or hypertensive encephalopathy
* abdominal fistula, gastrointestinal bleeding, or intra-abdominal abscess within the 6 months prior to study enrollment.
* core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment.
* major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study.
* recent arterial thrombotic events including stroke or TIA within 6 months prior to study enrollment.
* serious or non-healing wound, ulcer or bone fracture.
* active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-05; Primary Completion 2013-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Lacy, M.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Medical Oncology & Hematology PC, Hamden, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFOX/Bevacizumab Administration: FOLFOX in combination with bevacizumab
  FOLFOX: Oxaliplatin 85/mg/m2 IV infused over two hours followed by Leucovorin 400 mg/m2 IV over 2 hours, followed by 5-FU 400 mg/m2 IV bolus, then 2400 mg/m2 continuous IV infusion over 46-48 hours
  bevacizumab: bevacizumab will be used at a dose of 10 mg/kg administered every 2 weeks on day one of FOLFOX chemotherapy
Period: Overall Study
Arm/Group | FOLFOX/Bevacizumab Administration
Started | 39
Completed | 3
Not Completed | 36
Not completed — Progressive disease | 27
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 3
Not completed — Investigators' discretion | 2

BASELINE CHARACTERISTICS:
Arm/Group | FOLFOX/Bevacizumab Administration
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 62 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Time Frame: Upon completion of study, up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOX/Bevacizumab Administration
Number analyzed (Participants) | 39
months | 7.8 [5.9 to 11.6]

2. Secondary Outcome: Overall Tumor Response Rate by RECIST Criteria
Description: Per response evaulation criteria in solid tumors criteria (RECIST) for target lesions assessed by FDG-PET Scans: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: Upon completion of study
Measure: Number; unit: percentage of participants
Arm/Group | FOLFOX/Bevacizumab Administration
Number analyzed (Participants) | 39
percentage of participants | 56.4

3. Secondary Outcome: Overall Survival
Time Frame: Upon completion of study, up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOX/Bevacizumab Administration
Number analyzed (Participants) | 39
months | 14.7 [11.5 to 16.6]

ADVERSE EVENTS:
Time Frame: Toxicity assessment were performed up to 3 years
Arm/Group | FOLFOX/Bevacizumab Administration
Serious Adverse Events (participants affected / at risk) | 4/39
Other Adverse Events (participants affected / at risk) | 16/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOX/Bevacizumab Administration (N=39)
Thromboytopenia (Blood and lymphatic system disorders) | 2
Neuropathy (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOX/Bevacizumab Administration (N=39)
Anemia (Blood and lymphatic system disorders) | 1
Neurtropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Fatigue (General disorders) | 3
Mucositis (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 4
Hand-Foot Syndrome (Skin and subcutaneous tissue disorders) | 1
Abnormal Liver Function Tests (Hepatobiliary disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Neuropathy (Nervous system disorders) | 8
Electrolytes Imbalence (General disorders) | 2
Deep Vein Thrombosis/Pulmonary Embolism (Vascular disorders) | 3
Hypertension (Vascular disorders) | 1
Proteinuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes